CLINICAL TRIAL: NCT02088372
Title: Evaluate Clinical Performance of Vanguard Knee With E1 Bearing in Korean Patient Population
Brief Title: Prospective Multi-Center Study on Vanguard With E1 Bearing
Acronym: VGRDE1
Status: Terminated | Type: Observational
Why Stopped: All 4 sites were terminated due to low follow-up of patients and low interest in the study
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: INT.CR.GK4
Record Dates: First submitted 2014-03-13; First posted 2014-03-14 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Varus Deformity; Valgus Deformity; Posttraumatic Deformity; Osteoarthritis, Knee; Unspecified Disorder of Knee Joint
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vanguard with E1 PS Bearing: E1™ Vitamin E doping of highly cross-linked polyethylene is a proposed method for insuring long-term oxidative stability of highly cross-linked ultra-high molecular weight polyethylene for use in total joint arthroplasty.
  Vanguard Total Knee System™ The Vanguard™ Knee System was designed to incorporate features from prior designs, including: ACG, Maxim, & Ascent.
  Interventions: Device: Vanguard with E1 PS Bearing

INTERVENTIONS:
Device: Vanguard with E1 PS Bearing — Evaluate Clinical Performance of Vanguard Knee with E1 Bearing in Korean Patient Population

SUMMARY:
Evaluate Clinical Performance of Vanguard Knee with E1 Bearing in Korean Patient Population

DETAILED DESCRIPTION:
E1™ Vitamin E doping of highly cross-linked polyethylene is a proposed method for insuring long-term oxidative stability of highly cross-linked ultra-high molecular weight polyethylene for use in total joint arthroplasty. In vitro research and development studies have shown that this material has improved wear performance, retention of mechanical properties, and a high resistance to oxidation due to the anti-oxidative properties of Vitamin E. Biomet Inc, has received FDA clearance to market tibial polyethylene components made of E1™ for use in the Vanguard total knee replacement system.

Vanguard Total Knee System™ The Vanguard™ Knee System was designed to incorporate features from prior designs, including: ACG, Maxim, & Ascent. The Vanguard Knee includes a streamlined design, rounded sagittal profile, and a deeper trochlear groove. The femoral component is available in Cruciate Retaining (CR), Posterior Stabilizing (PS), and Super Stabilized (SSK). Tibial Bearings are available in various levels of constraint required by the surgeon (CR, PS, AS, etc.).

For this study, ONLY Vanguard with PS Bearing will be used.

The purpose of the study is to evaluate clinical performance of Vanguard Knee with E1 Bearing in TKA in Korean patient population. The clinical performance will be evaluated based on patient outcomes, radiographic assessment and survivorship.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study if they received Vanguard knee with E1 Bearing per the approved indications for use for Vanguard Knee. Specifically

* Painful and disabled knee joint resulting from osteoarthritis or traumatic arthritis where one or more compartments are involved
* Correction of varus, valgus, or posttraumatic deformity
* Correction or revision of unsuccessful osteotomy

Exclusion Criteria:

Exclusion Criteria for this study should comply with the stated contraindications on package inserts of Vanguard™ Knee and the E1™ Tibial Bearing. These indications are stated below:

Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Painful and disabled knee joint resulting from osteoarthritis or traumatic arthritis where one or more compartments are involved, varus, valgus, or posttraumatic deformity, and revision of unsuccessful osteotomy at Chungnam Nat'l Univ. Hospital, Kangwon Nat'l Univ. Hospital, Gacheon Uni. Gil Medical Center, and Chonbuk Nat'l Univ. Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 1 year
  scoring system to rate the knee and patient's functional abilities such as walking and stair climbing before and after TKA

SECONDARY OUTCOMES:
Knee Sociey Score | 6 Months
  scoring system to rate the knee and patient's functional abilities such as walking and stair climbing before and after TKA
Knee Society Score | 3 Years
  scoring system to rate the knee and patient's functional abilities such as walking and stair climbing before and after TKA
Knee Society Score | 5 Years
  scoring system to rate the knee and patient's functional abilities such as walking and stair climbing before and after TKA
KOOS | 6 Months
  Knee injuries & Osteoarthritis Outcome Score
KOOS | 1 Year
  Knee injuries & Osteoarthritis Outcome Score
KOOS | 3 Years
  Knee injuries & Osteoarthritis Outcome Score
KOOS | 5 Years
  Knee injuries & Osteoarthritis Outcome Score
EQ5D | 6 Months
  standardised instrument for use as a measure of health outcome.
EQ5D | 1 Year
  standardised instrument for use as a measure of health outcome.
EQ5D | 3 Years
  standardised instrument for use as a measure of health outcome.
EQ5D | 5 Years
  standardised instrument for use as a measure of health outcome.
Modified University of California Los Angeles (UCLA) Activity Score | 6 Months
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Modified University of California Los Angeles (UCLA) Activity Score | 1 Year
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Modified University of California Los Angeles (UCLA) Activity Score | 3 Years
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Modified University of California Los Angeles (UCLA) Activity Score | 5 Years
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Radiographic Assessment | Immediate Post-op(2 - 4 Weeks)
  Radiographic Evaluation
Radiographic Assessment | 6 Months
  Radiographic Evaluation
Radiographic Assessment | 1 Year
  Radiographic Evaluation
Radiographic Assessment | 3 Years
  Radiographic Evaluation
Radiographic Assessment | 5 Years
  Radiographic Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Young Mo Kim, Ph.D, Principal Investigator — Chungnam Nat'l Univ. Hospital; Kye Young Han, Ph.D, Principal Investigator — Kangwon Nat'l Univ. Hospital; Jae Ang Shim, Ph.D, Principal Investigator — Gacheon Uni. Gil Medical Center; Joo Hong Lee, Ph. D, Principal Investigator — Chonbuk Nat'l Univ. Hospital
Locations (4):
- South Korea (4):
  - Kangwon Nat'l Univ. Hospital, Chuncheon
  - Chungnam Nat'l Univ. Hospital, Daejeon
  - Gacheon Gil Univ. Gil Medical Center, Incheon
  - Chonbuk Nat'l Univ. Hospital, Jeonju

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2013-02-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02088372/Prot_000.pdf